CLINICAL TRIAL: NCT00758277
Title: Efficacy and Safety of Levetiracetam in Prevention of Alcohol Relapse in Recently Detoxified Alcohol Dependent Patients
Acronym: Keppra-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Martin Schaefer, MD, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Kep-F10.2.01
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Last update posted 2011-06-23 (Estimated); Status verified 2009-08

CONDITIONS: Alcohol Dependence; Alcoholic Relapse
Keywords: prevention of alcohol relapse
MeSH Terms: conditions — Alcoholism | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levetiracetam (Active Comparator)
  Interventions: Drug: levetiracetam (Keppra)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: levetiracetam (Keppra) — levetiracetam daily application 1500-2000 mg
  Other Names: KEPPRA
  Arms: Levetiracetam
Drug: Placebo — Sugar Pill
  Arms: Placebo

SUMMARY:
Prospective randomized double blind controlled trial in prevention of relapse in recently detoxified alcohol dependent patients with levetiracetam and placebo.

DETAILED DESCRIPTION:
Out-patients with alcohol dependence recently detoxified Primary goal size is the duration of the Abstinenz up to the heavy relapse.

Secondary objective size are:

* Frequency of Lapses
* Time up to the first alcohol drinking
* cumulative times of do not drink
* Craving
* Alcohol drinking quantity
* Sleep quality
* Tolerability/Bearableness of the study medication
* Security
* Drop Out rate
* Side effects
* Changes with the neuropsychological testing HAM-A, HAM-D, SF12, PSQI, VASC, OCDS, TLFB, SCL-90.
* Quality of life

ELIGIBILITY:
Inclusion Criteria:

* At least 18 and not older than 70 years
* Good knowledge of the German language
* The criteria of an alcohol dependence after DSM IV and ICD 10 fulfill
* To the recruiting time alkoholabstinently living, i.e. after successful alcohol decontamination, the patients must have understood the meaning and consequence of the study and have delivered before beginning of study your written agreement to the participation.
* Negative drug screening regarding Benzodiazepines and Opiates.
* With Females either o at least 1 year Menopause or after Sterilization or contraceptive pill, mini pill, three-monthly syringe, Implanton, Vaginalring, hormone plaster, hormone spiral at least 1 month before study inclusion or use of the double barrier method with Spermiziddiaphragma plus condom use or renouncement of sexual intercourse during the entire study duration and resolution a pregnancy to avoid with negative β-HCG-test

Exclusion Criteria:

* Alcohol withdrawal syndrome beginning or existing
* Simultaneous one ambulatory or stationary curing therapy, not however participation in groups of self-helps
* Specific ones behavior or deep-psychological single therapy or manual-led group therapies parallel to the clinical study
* Any further substance dependence except nicotine and/or Caffeine dependence A abuse according to the criteria of DSM-IV and/or ICD-10 is not considered as exclusion reason.
* Idiopathic epilepsy, not however admitted alcohol withdrawal convulsions
* Anamnesis of heavy cerebral traumas or other heavy neurological illnesses, not however alcohol-associated neurological disturbances, e.g. Polyneuropathie
* current CO-medication by means of medicines, which can affect significantly withdrawal symptoms or Craving or promote the Abstinent( Benzodiazepines, Antiepileptics, antipsychotics, Clonidin, antidepressives or Naltrexon (or substances with comparable effect mechanism) or Acamprosat, Disulfiram, or further substances, which can affect glutamaterge, dopaminerge, cholinergic, serotonerge or opiode system the GABAerge,
* Contraindications or heavy side effects in relation to the study medication, hypersensitivity opposite Pyrrolidonderivate
* Pregnancy or quiet time or insufficient Contraception
* Acute severe psychiatric disturbances in need of treatment of the axle I after DSM-IV
* Acute Suizidalität, not convincingly arrangementable
* Severe internal illnesses, e.g. Pancreatitis, pneumonia, cardiac infarct, gastrointestinal bleedings etc.)
* Severe kidney damage (starting from dekompensierter retention - stage 3 after that national Kidney Foundation) or heavy liver damage (starting from Child A after Child Pugh Score with living ore erring trousers) and/or creatinin Clearance of small 30ml/min
* Simultaneous participation or within the last 4 weeks at another clinical study, however does not exist an exclusion with previous participation in the decontamination study with Keppra ® (Keppra 1).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Comparison alcohol free "surviving "(heavy alcohol relapse) between experimental therapy (Keppra®) and a group of placebos | During and after treatment

SECONDARY OUTCOMES:
1 Time up to first drinking | During treatment
2 cumulative Time of do not drinking over the study duration | during treatment
3 Frequency of Lapses | during treatment
Tolerability of the study medication | during treatment
Drop Out rate | during treatment
Side effects | during treatment
Changes with the neuropsychological testing, HAM-A, HAM-D, SF12, VASC, OCDS, TLFB, SCL-90 | during treatment
Quality of life | during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Martin Schaefer, MD, Principal Investigator — Department of Psychiarty, Charite Campus Mitte, Berlin, and Department of Psychiatry, Kliniken Essen-Mitte, Essen, Germany
Locations (11):
- Germany (11):
  - Klinikum Nürnberg Nord, Nuremberg, Bavaria
  - Westfälisches Zentrum Bochum, Psychiatrie, Psychotherapie & Psychosomatik, Klinik der Ruhr-Universität, Bochum, North Rhine-Westphalia
  - Klinik und Poliklinik für Psychiatrie und Psychotherapie, Bonn, North Rhine-Westphalia
  - Klinik für Psychiatrie, Psychotherapie und Suchtmedizin Kliniken Essen - Mitte, Essen, North Rhine-Westphalia
  - Klinik für abhängiges Verhalten und Suchtmedizin, Rheinische Kliniken Essen, Kliniken der Universität Duisburg-Essen, Essen, North Rhine-Westphalia
  - Klinik für abhängiges Verhalten und Suchtmedizin, Rheinische Kliniken, Essen, Kliniken der Universität Duisburg - Essen, Essen, North Rhine-Westphalia
  - Klinik für Psychiatrie und Psychotherapie der Martin-Luther-Universität Halle, Halle, Saxony-Anhalt
  - Charité Campus Mitte, Klinik für Psychiatrie und Psychotherapie, Berlin, State of Berlin
  - PUK Charité im SHK, Berlin, State of Berlin
  - Vivantes, Wenckebach-Krankenhaus, Klinik für Psychiatrie und Psychotherapie, Gerontopsychiatrie/Psychosomatik, Berlin, State of Berlin
  - Klinik für Psychiatrie und Psychotherapie, Jüdisches Krankenhaus Berlin, Berlin, State of Berlin

REFERENCES:
- [Background] Krebs M, Leopold K, Richter C, Kienast T, Hinzpeter A, Heinz A, Schaefer M. Levetiracetam for the treatment of alcohol withdrawal syndrome: an open-label pilot trial. J Clin Psychopharmacol. 2006 Jun;26(3):347-9. doi: 10.1097/01.jcp.0000219926.49799.89. No abstract available. PMID 16702910
- [Derived] Richter C, Effenberger S, Bschor T, Bonnet U, Haasen C, Preuss UW, Heinz A, Forg A, Volkmar K, Glauner T, Schaefer M. Efficacy and safety of levetiracetam for the prevention of alcohol relapse in recently detoxified alcohol-dependent patients: a randomized trial. J Clin Psychopharmacol. 2012 Aug;32(4):558-62. doi: 10.1097/JCP.0b013e31825e213e. PMID 22722516